CLINICAL TRIAL: NCT02572479
Title: Observational Study for Evaluating the Potential of Diet and Food Components as Disease Modifiers in Amyotrophic Lateral Sclerosis (JERN_ALS)
Brief Title: Evaluating the Potential of the Diet as Disease Modifier in Amyotrophic Lateral Sclerosis (JERN_ALS)
Acronym: JERN_ALS
Status: Completed | Type: Observational
Sponsor: University of Jena (Other)
Collaborators: Jena University Hospital (Other)
Responsible Party: Principal Investigator, Christine Dawczynski,PhD, PhD, University of Jena
Other Study IDs: H01_15
Record Dates: First submitted 2015-10-06; First posted 2015-10-09 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2015-09

CONDITIONS: Amyotrophic Lateral Sclerosis; Dietary Habits; Disorder of Fatty Acid Metabolism
Keywords: fatty acids, amyotrophic lateral sclerosis, nutrient status
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sampling every six months (1x 9mL Sarstedt monovette)
Oversight: Data Monitoring Committee: No

SUMMARY:
The proposed observational trial will collect substantial data concerning dietary intake documented by ALS patients complemented by the analysis of fatty acid distribution in erythrocyte lipids. Both data sets are related to disease status and progress.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a currently incurable, multifactorial motor neuron disease characterized by upper and lower motor neuron degeneration, skeletal muscle atrophy, paralysis, and death. Multiple mechanisms caused by genetic and environmental factors proposed as responsible for ALS pathogenesis include decreased availability to neurotrophic factors, disturbances in calcium metabolism, increased neuroinflammatory status, cytoskeletal changes, mitochondrial dysfunction, dysfunction of protein degradation, glutamate excitotoxicity, apoptosis and oxidative stress.

Currently, the only available drug to treat ALS is riluzole which slightly prolongs life. Nutritional management has become more important in the treatment of ALS because body mass index and nutritional status seems to be independent, prognostic factors for survival and disease complications. Malnutrition is common in ALS, so caloric supplementation is essential. Additionally, many ALS patients self-medicate with vitamins, herbs, and other dietary supplements.

The objective of the current project is establishing the link between nutritional intake and disease status and progress. In detail, we like to assess if the improved outcomes are associated with specific nutrients, or simply the provision of excess calories. In this context, one of the most promising dietary candidates are polyunsaturated fatty acids (PUFA) and in particular the long-chain n-3 PUFA docosahexaenoic acid. This important structural component in neuronal membranes plays a role in neurogenesis and neuroprotection as well as exerts well-described anti-inflammatory effects in the brain.

The proposed observational trial will collect substantial data concerning dietary intake documented by ALS patients (Food Frequency Protocols, FFPs, periodic over 5 days) combined with the analysis of fatty acid distribution in erythrocyte lipids which reflects fatty acid distribution of the consumed fatty or oily foods (time period: approximately the last 2-3 months).

The fatty aids distribution in erythrocyte lipids as well as the nutrient intake calculated by FFPs are related to disease status and progress.

Thus, the current research activities focus on identification of dietary factors that are associated with disease progress or survival to develop beneficial interventions and therapy options.

ELIGIBILITY:
Inclusion Criteria:

* ALS patients diagnosed according to El Escorial / Awaji criteria for ALS
* patients should have the ability to comprehend the full nature and purpose of the study, to cooperate with the investigator, to understand verbal and written instructions, and to comply with the requirements of the entire study.

Exclusion Criteria:

* patient's request or if patient compliance with the study protocol is doubtful

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALS patients diagnosed according to El Escorial / Awaji criteria for ALS
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Clinical neurological examination | through study completion, an average of 1 year
  ALS functional rating scale-revised (ALSFRS-R)
  - the parameter will be assessed every three months through study completion

SECONDARY OUTCOMES:
Nutrient intake by diet | through study completion, an average of 1 year
  Food Frequency Protocol (FFP) over 5 days before blood sampling (FFP originate from Prodi® 6.4 software; Nutri-Science GmbH, Freiburg, Germany).
  Data analysis via Prodi®
  * calculation food nutrient profiles originated from the 'Bundeslebensmittelschlüssel'
  * calculation of daily energy intake, intake of fat and fatty acids, carbohydrates (individual sugars, dietary fibres), protein and amino acids, vitamins and minerals, sterols, etc.
  * the parameter will be assessed every three months through study completion
Fatty acid distribution in erythrocyte lipids | through study completion, an average of 1 year
  * marker for the fatty acid distribution of the consumed fatty or oily foods
  * reflect the fatty acid distribution of the consumed fatty or oily foods over the last 2-3 months as well as the endogenous metabolism and conversion of fatty acids
  * the parameter will be assessed every six months through study completion
Blood lipids | through study completion, an average of 1 year
  Total cholesterol, HDL-cholesterol, LCL-cholesterol, triacylglycerides
  - the parameter will be assessed every six months through study completion
Inflammatory parameter | through study completion, an average of 1 year
  c-reactive protein
  - the parameter will be assessed every six months through study completion
Metabolic serum parameters | through study completion, an average of 1 year
  glycated hemoglobin HbA1C
  - the parameter will be assessed every six months through study completion
Clinical neurological examination, part II | through study completion, an average of 1 year
  EQ5D-5L (population based QoL questionnaire)
  - the parameter will be assessed every six months through study completion

CONTACTS AND LOCATIONS:
Overall Officials: Julian Grosskreutz, PhD, Principal Investigator — Jena University Hospital, Hans Berger Department of Neurology; Christine Dawczynski, PhD, Principal Investigator — University of Jena, Department of Nutritional Biochemistry and Physiology; Stefan Lorkowski, Professor, Principal Investigator — University of Jena, Department of Nutritional Biochemistry and Physiology
Locations (1):
- Jena University Hospital, Hans Berger Department of Neurology, Jena, Thuringia, Germany